CLINICAL TRIAL: NCT03697252
Title: A Phase 2, Randomized, Double-blinded Study to Assess the Safety, Tolerability, and Efficacy of KarXT in Hospitalized Adults With DSM-5 Schizophrenia
Brief Title: A Study to Assess Safety and Efficacy of KarXT in Adult Patients With Schizophrenia
Acronym: EMERGENT-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karuna Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KAR-004
Record Dates: First submitted 2018-10-03; First posted 2018-10-05 (Actual); Results first posted 2020-09-28 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — xanomeline; trospium chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KarXT (Experimental)
  Interventions: Drug: Xanomeline and Trospium Chloride Capsules
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Capsules

INTERVENTIONS:
Drug: Xanomeline and Trospium Chloride Capsules — Xanomeline 50 mg/trospium 20 mg BID on days 1-2 followed by xanomeline 100 mg/trospium 20 mg BID on days 3-7. The dose is increased to xanomeline 125 mg/trospium 30 mg BID on days 8-34 unless the subject is experiencing adverse events from the xanomeline 100 mg/trospium 20 mg dose. Subjects who were increased to xanomeline 125 mg/trospium 30 mg will have the option to return to xanomeline 100 mg/trospium 20 mg depending on clinical response and tolerability. Dosing must not change after Visit 7 of the study (at 21 ± 2 days of dosing) and may be decreased for tolerability reasons no more than once during the study.
  Other Names: KarXT
  Arms: KarXT
Drug: Placebo Capsules — Placebo Capsules
  Arms: Placebo

SUMMARY:
This is a Phase 2, randomized, double-blinded, placebo-controlled, inpatient study to examine the efficacy, safety, and tolerability profile of KarXT in adult subjects diagnosed with DSM-5 schizophrenia who are in an acute exacerbation phase. The primary objective of the study is to assess the efficacy of KarXT (a fixed combination of xanomeline and trospium chloride) (xanomeline 125 mg/trospium 30 mg twice daily [BID]) versus placebo in reducing Positive and Negative Syndrome Scale (PANSS) total scores in adult inpatients with a Diagnostic and Statistical Manual-Fifth Edition (DSM-5) diagnosis of schizophrenia. The secondary objectives of the study are to assess overall safety and tolerability of KarXT in adult inpatients with a DSM-5 diagnosis of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is aged 18-60 years, inclusive, at screening
2. Subject has a primary diagnosis of schizophrenia established by a comprehensive psychiatric evaluation based on the DSM-5 (American Psychiatric Association 2013) criteria and confirmed by Mini International Neuropsychiatric Interview for Schizophrenia and Psychotic Disorder Studies (MINI) version 7.0.2.
3. Subject is experiencing an acute exacerbation or relapse of symptoms, with onset less than 2 months before screening
4. Positive and Negative Syndrome Scale total score between 80 and 120, inclusive, at screening

   1. Score of ≥ 4 (moderate or greater) for ≥ 2 of the following Positive Scale (P) items at screening:
   2. Item 1 (P1; delusions)
   3. Item 2 (P2; conceptual disorganization)
   4. Item 3 (P3; hallucinatory behavior)
   5. Item 6 (P6; suspiciousness/persecution)
5. There should not be a change (improvement) in PANSS total score between screening and baseline of more than 20%
6. Subjects taking a depot antipsychotic could not have received a dose of medication for at least 1 and a half injection cycles before baseline (eg, 3 or more weeks off for a 2-week cycle)
7. Subject is capable of providing informed consent

   1. A signed ICF must be provided before any study assessments are performed
   2. Subject must be fluent (oral and written) in English in order to consent
8. Subject must have CGI-S score of ≥ 4 at screening and baseline visits
9. Body mass index must be ≥ 18 and ≤ 40 kg/m2
10. Both females of child bearing potential and males with partners of child bearing potential must be willing to use a double-barrier method of birth control (ie, any double combination of male or female condom with spermicidal gel, diaphragm, sponge, or cervical cap with spermicidal gel) during the study and for 7 days after the last dose of study drug.
11. Subject has an identified reliable informant

Exclusion Criteria:

1. Any primary DSM-5 disorder other than schizophrenia within 12 months before screening (confirmed using MINI version 7.0.2 at screening)
2. History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or oncologic disease or any other condition that, in the opinion of the investigator, would jeopardize the safety of the subject or the validity of the study results, to exclude patients with human immunodeficiency virus (HIV), cirrhosis, biliary duct abnormalities, hepatobiliary carcinoma, and/or active hepatic viral infections based on the liver function test results.
3. History of or high risk of urinary retention, gastric retention, or narrow-angle glaucoma
4. History of irritable bowel syndrome (with or without constipation) or serious constipation requiring treatment within the last 6 months
5. Has a DSM-5 diagnosis of moderate to severe substance abuse disorder (except tobacco use disorder) within the 12 months before screening (confirmed using MINI version 7.0.2 at screening), or current abuse as determined by urine toxicology screen or alcohol test. A screening subject with mild substance abuse disorder within the 12 months before screening must be discussed and agreed upon with the medical monitor before he/she can be allowed into the study.
6. Clinically significant abnormal finding on the physical examination, medical history, ECG, or clinical laboratory results at screening
7. Pregnant, lactating, or less than 3 months postpartum. Sperm donation is not allowed for 90 days after the final dose of study drug
8. If, in the opinion of the investigator (and/or Sponsor), subject is unsuitable for enrollment in the study or subject has any finding that, in the view of the investigator (and/or Sponsor), may compromise the safety of the subject or affect their ability to adhere to the protocol visit schedule or fulfill visit requirements
9. Subject has had psychiatric hospitalization(s) for more than 30 days (cumulative) during the 90 days before screening
10. Subject has a history of treatment resistance to schizophrenia medications defined as failure to respond to 2 adequate courses of pharmacotherapy (a minimum of 4 weeks at an adequate dose per the label) or required clozapine within the last 12 months
11. Risk of violent or destructive behavior
12. Current involuntary hospitalization or incarceration
13. Participation in another clinical study in which the subject received an experimental or investigational drug agent within 3 months of screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 182 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2019-09-04 (Actual); Study Completion 2019-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Brannan, MD, Study Director — Karuna Therapeutics
Locations (12):
- United States (12):
  - Woodland International Research Group, LLC, Little Rock, Arkansas
  - Synergy East, Lemon Grove, California
  - Collaborative Neuroscience Network, LLC., Long Beach, California
  - NRC Research Institute, Orange, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - CBH Health, LLC, Gaithersburg, Maryland
  - Hassman Research Institute, Berlin, New Jersey
  - Midwest Clinical Research Center (and IP Shipment), Dayton, Ohio
  - Community Clinical Research, Inc., Austin, Texas
  - InSite Clinical Research, LLC, DeSoto, Texas
  - Pillar Clinical Research, LLC, Richardson, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yeung PP, Breier A, Zhu H, Kaul I, Marcus RN. Xanomeline and Trospium Chloride for the Treatment of Agitation Associated With Schizophrenia: PANSS-Excited Component Results From 3 Randomized, Double-Blind, Placebo-Controlled EMERGENT Trials. J Clin Psychiatry. 2025 Mar 24;86(2):24m15668. doi: 10.4088/JCP.24m15668. PMID 40215379
- [Derived] Citrome L, Neugebauer NM, Meli AA, Kando J. Xanomeline and Trospium Chloride Versus Placebo for the Treatment of Schizophrenia: A Post Hoc Analysis of Number Needed to Treat, Number Needed to Harm, and Likelihood to Be Helped or Harmed. Neuropsychiatr Dis Treat. 2025 Apr 5;21:761-773. doi: 10.2147/NDT.S503494. eCollection 2025. PMID 40212458
- [Derived] Kaul I, Claxton A, Sawchak S, Sauder C, Brannan SK, Raj E, Ruan S, Konis G, Brown D, Cutler AJ, Marcus R. Safety and Tolerability of Xanomeline and Trospium Chloride in Schizophrenia: Pooled Results From the 5-Week, Randomized, Double-Blind, Placebo-Controlled EMERGENT Trials. J Clin Psychiatry. 2025 Feb 26;86(1):24m15497. doi: 10.4088/JCP.24m15497. PMID 40047530
- [Derived] Sauder C, Allen LA, Baker E, Miller AC, Paul SM, Brannan SK. Effectiveness of KarXT (xanomeline-trospium) for cognitive impairment in schizophrenia: post hoc analyses from a randomised, double-blind, placebo-controlled phase 2 study. Transl Psychiatry. 2022 Nov 21;12(1):491. doi: 10.1038/s41398-022-02254-9. PMID 36414626
- [Derived] Weiden PJ, Breier A, Kavanagh S, Miller AC, Brannan SK, Paul SM. Antipsychotic Efficacy of KarXT (Xanomeline-Trospium): Post Hoc Analysis of Positive and Negative Syndrome Scale Categorical Response Rates, Time Course of Response, and Symptom Domains of Response in a Phase 2 Study. J Clin Psychiatry. 2022 May 11;83(3):21m14316. doi: 10.4088/JCP.21m14316. PMID 35552528
- [Derived] Targum SD, Murphy C, Breier A, Brannan SK. Site-independent confirmation of primary site-based PANSS ratings in a schizophrenia trial. J Psychiatr Res. 2021 Dec;144:241-246. doi: 10.1016/j.jpsychires.2021.10.027. Epub 2021 Oct 21. PMID 34700212
- [Derived] Brannan SK, Sawchak S, Miller AC, Lieberman JA, Paul SM, Breier A. Muscarinic Cholinergic Receptor Agonist and Peripheral Antagonist for Schizophrenia. N Engl J Med. 2021 Feb 25;384(8):717-726. doi: 10.1056/NEJMoa2017015. PMID 33626254

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 12 study centers in North America.
Pre-assignment Details: A total of 250 participants were screened, 182 were randomized, and 145 participants completed the study.
Groups:
- KarXT: Participants received oral Capsule KarXT (xanomeline 125 mg/trospium 30 mg BID) in a treatment period of 5 weeks. Participants were started on a lead in dose of xanomeline 50 mg/trospium 20 mg twice a day (BID) for the first 2 days followed by xanomeline 100 mg/trospium 20 mg BID for the remainder of Week 1 (Days 3 to 7). On Day 8, dosing was titrated upwards to xanomeline 125 mg/trospium 30 mg BID unless the Participant was continuing to experience adverse events from the previous dose increase of xanomeline 100 mg/trospium 20 mg BID. All Participants who were increased to xanomeline 125 mg/trospium 30 mg BID, depending on clinical response and tolerability, had the option to return to xanomeline 100 mg/trospium 20 mg BID for the remainder of the treatment period.
- Placebo: Participants received the matching placebo to KarXT orally twice daily for a treatment period of 5 weeks.
Period: Overall Study
Arm/Group | KarXT | Placebo
Started | 90 | 92
Completed | 72 | 73
Not Completed | 18 | 19
Not completed — Adverse Event | 3 | 2
Not completed — Withdrawal by Subject | 14 | 14
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) population included all participants who were randomized to the study. Participants were analyzed according to randomized treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | KarXT | Placebo | Total
Number analyzed (Participants) | 90 | 92 | 182
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.4 (10.12) | 41.6 (10.08) | 42.5 (10.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 24 | 42
  Male | 72 | 68 | 140
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 67 | 70 | 137
  White | 20 | 17 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at Week 5
Description: The PANSS is a medical scale used for measuring symptom severity of participants with schizophrenia. The PANSS rating form contains 7 positive symptom scales, 7 negative system scales, and 16 general psychopathology symptom scales. Participants were rated from 1 to 7 on each symptom scale. The total score is the sum of all scales with a minimum score of 30 and a maximum score of 210. A decrease in PANSS total score correlates with an improvement in schizophrenia symptoms.
Time Frame: Baseline and Week 5
Population: The Modified Intent-to-Treat (MITT) population included all participants who were randomized, received at least one dose of study medication, and had a baseline and at least one post-baseline PANSS assessment. Here, the number of participants analyzed indicates participants who were evaluable for this measure at given time points for each group.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 83 | 87
score on a scale | -17.40 (1.749) | -5.85 (1.668)
Statistical Analysis 1: Comparison: KarXT vs Placebo; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; LS mean difference = -11.56, 95% CI 2-sided [-16.07 to -7.05]; Statistics are from a mixed model for repeated measures (MMRM). The model includes the treatment group (KarXT or placebo), visit, and the interaction between the treatment group and visit as fixed factors, and baseline PANSS total score, site, age, and gender as covariates. An unstructured covariance matrix is used to model the correlation among repeated measurements and the denominator degrees of freedom are computed using the Kenward-Roger method

2. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Positive Score at Week 5
Description: The PANSS is a medical scale used for measuring symptom severity of participants with schizophrenia. The PANSS rating form contains 7 positive symptom scales, 7 negative system scales, and 16 general psychopathology symptom scales. The positive symptoms in schizophrenia are the excess or distortion of normal functions such as hallucinations, delusions, grandiosity, and hostility. Participants were rated from 1 to 7 on each symptom scale, with a minimum score of 7 and a maximum score of 49. A decrease in PANSS total score correlates with an improvement in schizophrenia symptoms.
Time Frame: Baseline and Week 5
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 83 | 87
score on a scale | -5.62 (0.601) | -2.38 (0.573)

3. Secondary Outcome: Number of Participants With Each Clinical Global Impression - Severity (CGI-S) Score at Baseline and 5 Weeks
Description: The CGI-S modified asked the clinician 1 question: "Considering your total clinical experience, how mentally ill is the participant at this time?" The clinician's answer rated on the following 7-point scale: 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; 7 = among the most extremely ill participants.
Time Frame: Baseline and Week 5
Population: The MITT population included all participants who were randomized, received at least one dose of study medication, and had a baseline and at least one post-baseline PANSS assessment. Here, the number of participants analyzed indicates participants who were evaluable for this measure at given time points for each group.
Measure: Count of Participants; unit: Participants
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 83 | 87
Participants
  Baseline: Score = 1 | 0 | 0
  Week 5: Score = 1: number analyzed (Participants) | 72 | 73
  Week 5: Score = 1 | 1 | 0
  Baseline: Score = 2 | 0 | 0
  Week 5: Score = 2: number analyzed (Participants) | 72 | 73
  Week 5: Score = 2 | 3 | 1
  Baseline: Score = 3 | 0 | 0
  Week 5: Score = 3: number analyzed (Participants) | 72 | 73
  Week 5: Score = 3 | 23 | 7
  Baseline: Score = 4 | 13 | 17
  Week 5: Score = 4: number analyzed (Participants) | 72 | 73
  Week 5: Score = 4 | 21 | 21
  Baseline: Score = 5 | 60 | 60
  Week 5: Score = 5: number analyzed (Participants) | 72 | 73
  Week 5: Score = 5 | 21 | 38
  Baseline: Score = 6 | 10 | 9
  Week 5: Score = 6: number analyzed (Participants) | 72 | 73
  Week 5: Score = 6 | 2 | 4
  Baseline: Score = 7 | 0 | 1
  Week 5: Score = 7: number analyzed (Participants) | 72 | 73
  Week 5: Score = 7 | 1 | 2
Statistical Analysis 1: Comparison: KarXT vs Placebo; Comparison of KarXT and Placebo at Week 5; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Negative Score at Week 5
Description: The PANSS is a medical scale used for measuring symptom severity of participants with schizophrenia. The PANSS rating form contains 7 positive symptom scales, 7 negative system scales, and 16 general psychopathology symptom scales. The negative symptoms in schizophrenia are the diminution or loss of normal functions. Participants were rated from 1 to 7 on each symptom scale, with a minimum score of 7 and a maximum score of 49. A decrease in PANSS total score correlates with an improvement in schizophrenia symptoms.
Time Frame: Baseline and Week 5
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 83 | 87
score on a scale | -3.18 (0.481) | -0.90 (0.454)

5. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Marder Factor Score
Description: The Marder Negative Factor score is derived from the PANSS and consists of the sum of 5 negative scales (N) and 2 general scales (G) (N1. Blunted affect; N2. Emotional withdrawal; N3. Poor rapport; N4. Passive/apathetic social withdrawal; N6. Lack of spontaneity; G7. Motor retardation; and G16. Active social avoidance), with a minimum score of 7 and a maximum score of 49.
Time Frame: Baseline and Week 5
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 83 | 87
score on a scale | -3.85 (0.520) | -1.32 (0.492)

6. Secondary Outcome: Percentage of Participants Who Were Clinical Global Impression - Severity of Illness (CGI-S) Responders
Description: The CGI-S modified asks the clinician 1 question: "Considering your total clinical experience, how mentally ill is the participant at this time?" The clinician's answer was rated on the following 7-point scale: 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; 7 = among the most extremely ill participants. A CGI-S responder is defined as a participant with a CGI-S scale equal to 1 or 2.
Time Frame: Week 5
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 72 | 73
percentage of participants | 5.6 | 1.4

ADVERSE EVENTS:
Time Frame: From the start of study drug administration up to Week 5
Description: The Safety population included all participants who received at least one dose of study medication.
Arm/Group | KarXT | Placebo
All-Cause Mortality (participants affected / at risk) | 0/89 | 0/90
Serious Adverse Events (participants affected / at risk) | 1/89 | 0/90
Other Adverse Events (participants affected / at risk) | 48/89 | 39/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KarXT (N=89) | Placebo (N=90)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KarXT (N=89) | Placebo (N=90)
Constipation (Gastrointestinal disorders) | 15 (16) | 3 (3)
Nausea (Gastrointestinal disorders) | 15 (15) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 8 (8) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 8 (11) | 4 (4)
Vomiting (Gastrointestinal disorders) | 8 (8) | 4 (4)
Headache (Nervous system disorders) | 6 (7) | 5 (5)
Somnolence (Nervous system disorders) | 5 (5) | 4 (4)
Akathisia (Nervous system disorders) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 3 (3)
Weight increased (Investigations) | 3 (3) | 4 (4)
Tachycardia (Cardiac disorders) | 3 (3) | 2 (2)
Sedation (Nervous system disorders) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 4 (4)
Gamma-Glutamyltransferase increased (Investigations) | 2 (2) | 0 (0)
Agitation (Psychiatric disorders) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-12-13): https://cdn.clinicaltrials.gov/large-docs/52/NCT03697252/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/52/NCT03697252/SAP_001.pdf